CLINICAL TRIAL: NCT00945854
Title: Effect of Whole Grain Rich Diet on Insulin Sensitivity in Individuals With Metabolic Syndrome
Brief Title: Wholegrain Cereal Diet and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, prof, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04022009; European Community
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-05

CONDITIONS: Metabolic Syndrome
Keywords: wholegrain cereals; glycemic index; metabolic syndrome; insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wholegrain cereal diet (Active Comparator): Treatment with a diet based on wholegrain cereals and foods with low glycemic index
  Interventions: Other: Wholegrain cereal diet
- Refined cereal diet (Active Comparator): Treatment with a diet based on refined cereals and foods with high glycemic index
  Interventions: Other: Refined cereal diet

INTERVENTIONS:
Other: Wholegrain cereal diet — Thirty subjects with metabolic syndrome, after an initial run-in period of 4 weeks, during which they stabilise their own diet and other lifestyle habits, are assigned to a diet based on wholegrain cereals and foods with low glycemic index for a period of 12 weeks. Before and after the dietary treatment, a frequently samples intravenous glucose tolerance is carried out to measure the effects of the intervention on glucose and insulin metabolism. At beginning and at the end of intervention, the subjects consume also a standard test meal to evaluate the postprandial response of glucose, insulin, lipids, oxidative parameters and inflammatory molecules.
  Arms: Wholegrain cereal diet
Other: Refined cereal diet — Thirty subjects with metabolic syndrome, after an initial run-in period of 4 weeks, during which they stabilise their own diet and other lifestyle habits, are assigned to a diet based on refined cereals and foods with high glycemic index for a period of 12 weeks. Before and after the dietary treatment, a frequently samples intravenous glucose tolerance is carried out to measure the effects of the intervention on glucose and insulin metabolism. At beginning and at the end of intervention, the subjects consume also a standard test meal to evaluate the postprandial response of glucose, insulin, lipids, oxidative parameters and inflammatory molecules.
  Arms: Refined cereal diet

SUMMARY:
A diet with the multiple beneficial characteristics of whole grains and, more in general, of "healthy cereals" favorably influences glucose and insulin metabolism in subjects with metabolic syndrome. Therefore, the aim of the study is to evaluate the long term effects of a diet containing "healthy cereals" versus a control diet, on glucose and insulin metabolism in subjects with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least three of the following criteria of metabolic syndrome according to ATPIII-NCEP criteria:

  1. waist circumference >102 for men and 88 for women,
  2. fasting total serum triacyglycerol concentration >1.7 mmol/L,
  3. fasting HDL cholesterol <1.0 mmol/L for men or <1.3 mmol/L for women,
  4. IFG (plasma glucose between 6.1 and 6.9 mmol/L) or
  5. blood pressure >130/85 mmHg or use of blood pressure medication
* Hypertension in stable control (BP <135/80 mmHg) by means of drugs, which will not be allowed to be changed during the study
* Absence of main cardiovascular events (IMA, Ictus)

Exclusion Criteria:

* Diabetes mellitus diagnosed according to history of diabetes or blood glucose ≥ 200 mg/dL (11.1 mmol/L) 2 hours after a 75 g Oral glucose tolerance test (OGTT) to be performed during the run-in period in all the subjects
* Any drug able to influence glucose and lipid metabolism (hypolipidemic drugs, cholesterol lowering foodstuffs, anti-inflammatory drugs)
* Renal failure (serum creatinine > 1.5 mg/dL) and liver failure (ALT/AST> 2 times above normal values)
* Anemia (Hb < 12g/dl) or any other chronic disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Riccardi, Prof., Study Chair — Dept. of Clinical and Experimental Medicine, Federico II University
Locations (1):
- Dept. of Clinical and Experimental Medicine, Federico II University, Naples, Italy

REFERENCES:
- [Background] Giacco R, Clemente G, Cipriano D, Luongo D, Viscovo D, Patti L, Di Marino L, Giacco A, Naviglio D, Bianchi MA, Ciati R, Brighenti F, Rivellese AA, Riccardi G. Effects of the regular consumption of wholemeal wheat foods on cardiovascular risk factors in healthy people. Nutr Metab Cardiovasc Dis. 2010 Mar;20(3):186-94. doi: 10.1016/j.numecd.2009.03.025. Epub 2009 Jun 7. PMID 19502018
- [Derived] Costabile G, Vetrani C, Bozzetto L, Giacco R, Bresciani L, Del Rio D, Vitale M, Della Pepa G, Brighenti F, Riccardi G, Rivellese AA, Annuzzi G. Plasma TMAO increase after healthy diets: results from 2 randomized controlled trials with dietary fish, polyphenols, and whole-grain cereals. Am J Clin Nutr. 2021 Oct 4;114(4):1342-1350. doi: 10.1093/ajcn/nqab188. PMID 34091663
- [Derived] Vitale M, Hanhineva K, Koistinen V, Auriola S, Paananen J, Costabile G, Della Pepa G, Rivellese AA, Riccardi G, Giacco R. Putative metabolites involved in the beneficial effects of wholegrain cereal: Nontargeted metabolite profiling approach. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1156-1165. doi: 10.1016/j.numecd.2020.12.022. Epub 2020 Dec 30. PMID 33589320
- [Derived] Polito R, Costabile G, Nigro E, Giacco R, Vetrani C, Anniballi G, Luongo D, Riccardi G, Daniele A, Annuzzi G. Nutritional factors influencing plasma adiponectin levels: results from a randomised controlled study with whole-grain cereals. Int J Food Sci Nutr. 2020 Jun;71(4):509-515. doi: 10.1080/09637486.2019.1680959. Epub 2019 Oct 22. PMID 31638838
- [Derived] Karkkainen O, Lankinen MA, Vitale M, Jokkala J, Leppanen J, Koistinen V, Lehtonen M, Giacco R, Rosa-Sibakov N, Micard V, Rivellese AAA, Schwab U, Mykkanen H, Uusitupa M, Kolehmainen M, Riccardi G, Poutanen K, Auriola S, Hanhineva K. Diets rich in whole grains increase betainized compounds associated with glucose metabolism. Am J Clin Nutr. 2018 Nov 1;108(5):971-979. doi: 10.1093/ajcn/nqy169. PMID 30256894

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wholegrain Cereal Diet | Refined Cereal Diet
Started | 30 | 30
Completed | 28 | 26
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wholegrain Cereal Diet | Refined Cereal Diet | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (8.5) | 57.4 (7.3) | 57.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity (Si)
Description: Peripheral insulin sensitivity was assessed by FSIGT. A glucose dose of 300 mg/kg body weight was given intravenously followed by a bolus of 0.03 U/kg of insulin injected after 20 min. Blood samples were frequently collected for 3 h for the measurement of plasma glucose and serum insulin concentrations, utilized to calculate the insulin sensitivity index Si
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: 104xmin-1/microU/ml
Arm/Group | Wholegrain Cereal Diet | Refined Cereal Diet
Number analyzed (Participants) | 28 | 26
104xmin-1/microU/ml | 3.03 (0.16) | 3.15 (0.19)
Statistical Analysis 1: Comparison: Wholegrain Cereal Diet vs Refined Cereal Diet; Test type: Superiority or Other; p < 0.05, ANCOVA

2. Secondary Outcome: Postprandial Insulin Changes
Description: Blood samples during the standard meal test were drawn from an antecubital vein after a 12 h overnight fast and 0, 30, 60, 90, 120, 150 and 180 min postprandial for the measurement of plasma insulin response reported as average mean postprandial increment.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: (microU/mlx3hrs)
Arm/Group | Wholegrain Cereal Diet | Refined Cereal Diet
Number analyzed (Participants) | 28 | 26
(microU/mlx3hrs) | 50.01 (10.2) | 64.4 (12.4)

3. Secondary Outcome: Postprandial Plasma Lipid Changes
Description: Blood samples during the standard meal test were drawn from an antecubital vein after a 12 h overnight fast and 0, 30, 60, 90, 120, 150 and 180 min postprandial for the measurement of triglyceride response reported as average mean postprandial increment.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dlx3hrs
Arm/Group | Wholegrain Cereal Diet | Refined Cereal Diet
Number analyzed (Participants) | 28 | 26
mg/dlx3hrs | 22.7 (4.2) | 47.6 (6.8)

ADVERSE EVENTS:
Arm/Group | Wholegrain Cereal Diet | Refined Cereal Diet
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No